CLINICAL TRIAL: NCT07263490
Title: PRIOR Study (Pre-eclampsia Risk In Oocyte Recipients) - Investigating Matching, Biomarkers and Outcomes.
Brief Title: PRIOR Study (Pre-eclampsia Risk In Oocyte Recipients)
Acronym: PRIOR
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Ferring Pharmaceuticals (Industry); Gedeon Richter Ltd. (Industry)
Responsible Party: Principal Investigator, Pernille Fog Svendsen, Associate Professor, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-22068878; p-2024-17237 (Registry Identifier: Privacy.legal)
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Pre-eclampsia; Oocyte Donation; Pre-Eclampsia; Complicating Pregnancy; Pre-Eclampsia; Mild; Pre-Eclampsia, Severe; Pre-eclampsia or Eclampsia With Pre-existing Hypertension; ART; Neonatal Morbidity; Neonatal Mortality; Placental Abruption; Gestational Diabetes; Preterm Labor; Post-partum Hemorrhage (PPH); Intrauterine Growth Restriction (IUGR); Hypertensive Disorders of Pregnancy
Keywords: Pre-eclampsia; Preeclampsia; ART; Gestational hypertension; Oocyte donation; Egg donation; Gamete donation
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Lymphoma, Follicular; Abruptio Placentae; Diabetes, Gestational; Obstetric Labor, Premature; Postpartum Hemorrhage; Fetal Growth Retardation; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples six times throughout the participants' pregnancies. Samples will be analyzed for pre-eclampsia markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preg OD: Women pregnant after treatment with oocyte donation
- Preg IVF: Women pregnant after IVF treatment with autologous oocytes

SUMMARY:
The aim of this prospective observational cohort study is to investigate the pathophysiological mechanisms behind and risk of pre-eclampsia in women pregnant after fertility treatment with oocyte donation. The participants are included in of of two cohorts. One includes women pregnant after oocyte donation whereas the other includes women pregnant after IVF treatment with autologous oocytes.

Participants will be followed throughout pregnancy with blood samples, blood pressure, clinical controls and ultrasound examinations. Clinical outcomes will be registered post-partum.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND Maternal age at conception has increased globally, leading to a higher proportion of pregnancies among women aged ≥35 years. In Denmark, the average maternal age at first birth has risen from 24 years in 1970 to 30 years in 2021. As female fecundity declines markedly after age 35, the need for assisted reproductive technology (ART) is increasing.

The success rate of ART using autologous oocytes decreases significantly after age 40, making oocyte donation (OD) a relevant option for women with diminished ovarian reserve or poor oocyte quality. OD was first introduced in 1984 to treat infertility due to premature ovarian failure and is now used for various indications including Turner syndrome, previous oophorectomy, gonadotoxic therapy, and certain genetic disorders.

OD has been legal in Denmark since 2007 and double gamete donation since 2018. Healthy women under 36 years can donate oocytes anonymously or non-anonymously. The number of OD procedures in Denmark has increased from 124 in 2011 to 2,782 in 2022, resulting in 756 deliveries in 2021. The rise is attributed to delayed motherhood, legal changes, and increased donor compensation.

Several studies have demonstrated that pregnancies following OD are associated with a higher risk of obstetric complications, including pre-eclampsia (PE), intrauterine growth restriction, preterm birth, cesarean section, placental abruption, and postpartum hemorrhage. The risk appears to be even higher in double gamete donation pregnancies. The mechanisms behind these associations remain unclear but are thought to involve immune maladaptation due to exposure to non-self paternal and donor antigens.

PE complicates approximately 3-8% of pregnancies and is defined as new-onset hypertension (≥140/90 mmHg) with proteinuria (≥300 mg/24 h) and/or signs of organ dysfunction after 20 weeks of gestation. Risk factors include prior PE, chronic hypertension, renal disease, diabetes, autoimmune disease, multifetal gestation, nulliparity, advanced maternal age, high BMI, long interpregnancy interval, and family history of PE.

PE and related disorders share a common pathophysiology involving abnormal placentation, impaired trophoblast invasion, and endothelial dysfunction. The etiology is multifactorial and may include genetic, immunological, and vascular components. Recent data indicate that fetal-maternal HLA mismatches, particularly HLA-DR incompatibility, are associated with increased PE risk.

This study hypothesizes that OD pregnancies, known to have elevated risk of PE, provide a relevant model to investigate the pathophysiological mechanisms of the disease.

STUDY OBJECTIVE The aim of this prospective observational cohort study is to investigate the pathophysiological mechanisms and the risk of pre-eclampsia in women who become pregnant following fertility treatment with oocyte donation.

The study population comprises two cohorts. These are a cohort of women pregnant after oocyte donation compared with a cohort of women pregnant after IVF with autologous gametes.

PRIMARY RESEARCH QUESTIONS

* To assess the risk of pre-eclampsia in pregnancies conceived after single or double gamete donation compared with pregnancies achieved using autologous gametes.
* To investigate immunological and angiogenic biomarkers, as well as HLA tissue-type markers, involved in the pathogenesis of pre-eclampsia.
* To evaluate obstetric and neonatal outcomes, including pre-eclampsia, gestational diabetes, preterm birth, placental abruption, intrauterine growth restriction, asphyxia, neonatal morbidity, and mortality among women pregnant after oocyte or double donation in Denmark.
* To establish a comprehensive database and biobank to facilitate future research, including long-term follow-up studies of children born following oocyte donation.

Participants will be monitored throughout pregnancy with serial blood sampling, blood pressure measurements, clinical assessments, and ultrasound examinations. Clinical outcomes will be recorded postpartum.

INCLUSION OF PATIENTS STUDY POPULATION

The study will include two cohorts:

1. Women who achieve pregnancy following oocyte or double gamete donation (OD cohort).
2. Women who achieve pregnancy following IVF treatment with their own (autologous) frozen-thawed blastocysts (IVF control cohort).

Recruitment and Identification of Participants

Participants will be identified early in pregnancy through two recruitment pathways:

1. Fertility Clinic Recruitment (Gestational Week 7-8)

   o Women attending an early pregnancy ultrasound after ART will breifly be informed about the study by fertility clinic staff.
   * If the woman expresses interest, her contact details (name, CPR number, and phone/email) will be forwarded to the principal investigator (PI).
   * The study team will contact the woman with detailed verbal and written information.
   * For women who are patients at Herlev Hospital, information will be provided in person, and a printed information sheet will be handed out.
   * For women treated at collaborating clinics (Rigshospitalet, Sellmer Fertility, Aleris Hamlet, Copenhagen Fertility Center, Trianglen), patient information will be provided via telephone, and written information will be either handed out or sent through secure digital mail (e-Boks).
2. Referral from General Practitioner (Gestational Week 8-10)

   o When women are referred from their general practitioner to the obstetric department, the visitation office will notify the PI of potential participants.
   * Written study information will be sent via secure e-mail (e-Boks), including notification that the woman will receive a phone call from study staff within a few days.
   * The woman will receive verbal information and may schedule an inclusion visit if interested.

   INFORMED CONSENT All participants will receive both verbal and written information about the study. Women will be encouraged to bring a companion or assessor to the inclusion visit. The inclusion visit includes repeated verbal information, opportunity for questions, and a minimum 24-hour reflection period before signing the consent form. Consent covers study participation, access to relevant clinical records, and collection of biological samples as specified in the protocol.

   ELIGIBILITY CRITERIA

   • Inclusion Criteria:

   o Pregnant women who conceived through oocyte donation, double gamete donation, or IVF treatment using their own (autologous) oocytes.

   o Ability to understand study information and provide written informed consent.

   o Willingness to participate in follow-up visits throughout pregnancy.

   • Exclusion Criteria:

   o Withdrawal of consent at any time during the study period.
   * Known multiple pregnancy at the time of inclusion.
   * Chronic medical conditions such as hypertension,

   INCLUSION Inclusion Visit (Gestational Week 10-12) (Visit 1) At the inclusion visit, informed consent will be obtained by the principal investigator or a trained study nurse. Eligibility criteria will be verified, and baseline data will be collected, including demographic information (age, ethnicity, family status), medical and fertility history, hereditary diseases, and current medication. Lifestyle factors such as smoking and alcohol use will be recorded.

   A physical examination will be performed, including height, weight, blood pressure, and heart rate. Routine fertility screening (smear, TSH, TPO, AMH, HIV, hepatitis, syphilis, rubella) will extracted from the patient files. Blood samples for study-specific analyses, including pre-eclampsia biomarkers, will be collected.

   Follow-up Visits (Visit 2-6 and telemedicine)

   Participants will undergo structured follow-up visits throughout pregnancy:

   • Gestational Week 12-14: Nuchal translucency ultrasound and blood sampling for pre-eclampsia markers.

   • Gestational Week 18-20: Detailed malformation ultrasound and blood sampling for pre-eclampsia markers.

   • Gestational Week 28: Initiation of weekly blood pressure measurements that are sent electronically to the hospital. Bloodsampling for pre-eclampsia markers.

   • Gestational Weeks 29-33: Weekly remote blood pressure monitoring sent to the hospital using an app.

   • Gestational Week 34: Clinical visit with ultrasound, obstetric examination, and blood sampling for pre-eclampsia markers. In addition remote blood pressure monitoring.
   * Gestational Weeks 35-37: Continued weekly remote blood pressure monitoring sent to the hospital using an app.
   * Gestational Week 38: Clinical visit with ultrasound, obstetric examination, and blood sampling for pre-eclampsia markers. In addition, remote blood pressure monitoring sent to the hospital using an app.
   * Gestational Week 39 until Delivery: Weekly remote blood pressure monitoring until delivery sent to the hospital using an app.

   Postpartum Data Collection After delivery, clinical outcome data will be obtained from electronic medical records. This includes gestational age at delivery, mode of delivery, birth weight, congenital malformations, and obstetric complications such as pre-eclampsia, gestational diabetes, intrauterine growth restriction, and postpartum hemorrhage.

   OUTCOME MEASURES

   Primary Outcome Measure:

   • Incidence of pre-eclampsia [Time Frame: From gestational week 20 until delivery]

   o Pre-eclampsia is defined as new-onset hypertension (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg) and proteinuria (≥300 mg/24h) and/or signs of organ dysfunction after 20 weeks of gestation. The primary outcome compares the incidence in pregnancies after oocyte or double gamete donation versus pregnancies after IVF with autologous oocytes.

   Secondary Outcome Measures:

<!-- -->

1. Immunological and angiogenic biomarkers [Time Frame: From inclusion until delivery]

   o Levels of specific biomarkers measured in maternal blood at multiple time points throughout pregnancy. Below are examples.

   o These are growth markers involved in early pregnancy (PAPP-A, IGF, PlGF, PGF and VEGFR), pro- and inflammatory cytokines (Interleukins, TNF-α and Interferon-γ), complement and thrombocyte activation markers (Selectin and BF-4), and markers for coagulation and fibrinolysis (Thrombin/anti-thrombin complexes and ex vivo fibrinogenesis/fibrinolysis).
2. HLA tissue type markers

   o Analysis of HLA mismatches between fetus and mother and their association with pre-eclampsia risk.
3. Obstetric complications [Time Frame: From inclusion until delivery]

   o Incidence of pre-eclampsia, postpartum hemorrhage, caesarean section, gestational diabetes, preterm birth (<37 weeks), IUGR, and placental abruption.
4. Neonatal outcomes [Time Frame: Birth until hospital discharge]

   * Incidence of intrauterine growth restriction, birth asphyxia, neonatal morbidity, and neonatal mortality.
5. Establishment of a database and biobank o Collection of clinical data and biological samples to enable future research, including potential long-term follow-up of children born after oocyte donation.

DATA COLLECTION AND HANDLING Signed informed consent allows access to relevant maternal and neonatal medical records for study purposes. All participant data will be collected in a secure electronic data capture system (REDCAP) compliant with local data protection regulations. Each participant will be assigned a unique study ID to ensure confidentiality. Source data will include electronic medical records, laboratory results, ultrasound reports, and telemedicine monitoring data. Only authorized study personnel will have access to identifiable data.

All study data will be recorded in case report forms (CRFs) and reviewed for completeness and accuracy. Queries will be resolved promptly with the study sites. Data will be backed up regularly, and audit trails will be maintained to track any changes to the dataset.

DATA STORAGE AND CONFIDENTIALITY Study data will be stored on secure servers with encryption. Access to identifiable information will be restricted to the principal investigator and designated study staff. Data will be retained for a minimum of 15 years following the end of the study, in accordance with institutional and national guidelines.

STATISTICAL ANALYSIS Data analysis will be performed according to a predefined statistical analysis plan. Descriptive statistics will be used to summarize baseline characteristics and clinical outcomes. Continuous variables will be expressed as means with standard deviations or medians with interquartile ranges, depending on distribution. Categorical variables will be presented as counts and percentages.

Comparisons between groups (e.g., oocyte donation vs. IVF pregnancies) will be conducted using appropriate statistical tests, such as t-tests or Mann-Whitney U tests for continuous variables and chi-square or Fisher's exact tests for categorical variables. Multivariable regression models will be applied to adjust for potential confounders.

All statistical tests will be two-sided, and a p-value <0.05 will be considered statistically significant. Interim analyses may be conducted if approved by the study steering committee, but final analyses will include all enrolled participants.

RISK MINIMIZATION The study involves minimal additional risk beyond standard clinical care for pregnant women. Blood draws will be performed by experienced personnel to minimize discomfort. Telemedicine monitoring will ensure timely detection of early signs of pre-eclampsia or other complications. Any participant developing severe complications will be referred for immediate clinical management according to standard obstetric protocols.

APPROVALS AND REGISTRATION The study is approved by the National Committee on Health Research Ethics (Approval no. H-22068878). This study was registered retrospectively on clinicaltrials.gov due to an administrative oversight in interpreting the prospective registration requirement. No changes were made to the protocol after study initiation. The research team has implemented revised internal procedures to ensure prospective registration for all future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* BMI < 35 kg/m2
* Normal wet smear within the past three years
* Both nulli- and multiparous
* Singletons and multiple gestations

Exclusion Criteria:

* Age < 18 years
* BMI > 35 kg/m2
* HIV/ hepatitis
* Essential hypertension
* Chronic kidney disease
* Undiagnosed vaginal bleeding
* Uterine malformations
* Persisting ovarian cysts
* Tumors in hypothalamus, pituitary, thyroid, or adrenal glands.
* Previous breast cancer
* Known BRCA 1 or 2 gene
* Unregulated thyroid disease
* Cardiovascular disease
* Breast feeding
* Present or previous chemotherapy/radiation therapy
* Present or previous malignant disease
* Smoking
* Alcohol/drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As this study explores risks during pregnancy and in delivery, the study is limited to persons with a uterus.
Study Population: Study population consists of women undergoing fertility treatment with IVF with either donated oocytes (Preg OD cohort) or autologous oocytes (Preg IVF cohort)
Sampling Method: Non-Probability Sample
Enrollment: 462 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Pre-eclampsia | During pregnancy and in the following two weeks post-partum
  Development of pre-eclampsia
Biochemical markers for pre-eclampsia | From early pregnancy untill delivery
  Analysis of bloodtests for biochemical markers of pre-eclampsia

SECONDARY OUTCOMES:
Post-partum hemorrhage | From delivery to 24 hours post-partum (Primary post-partum hemorrhage)
  Excessive bleeding (above 1000 mL) post-partum
Gestational diabetes | During pregnancy untill delivery.
Preterm delivery | Early delivery before gestational week 37
  Delivery before gestational week 37.
Placental abruption | During pregnancy and delivery
  Abruption of placenta
Intrauterine growth retardation (IUGR) | From pregnancy is obtained untill delivery
  Fetal growth restriction
Asphyxia | During delivery or in the first 24 hours post-partum
  Birth asphyxia
Neonatal morbidity | From delivery untill 28 days post-partum
  Presence of health complications or adverse outcomes in newborn during the first 28 days of life.
Neonatal mortality | From delivery untill 28 days post-partum
  Death of a live-born infant within 28 days of life

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Copenhagen Fertility Center, Copenhagen
  - Trianglen Fertility Clinic, Hellerup
  - Fertility Clinic, Herlev / Gentofte Hospital, Herlev
  - Sellmer Klinik, København S
  - Fertility Clinic, Rigshospitalet, København Ø
  - Aleris Fertility, Søborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian X, Aiyer KTS, Kapsenberg JM, Roelen DL, van der Hoorn ML, Eikmans M. Uncomplicated oocyte donation pregnancies display an elevated CD163-positive type 2 macrophage load in the decidua, which is associated with fetal-maternal HLA mismatches. Am J Reprod Immunol. 2022 Jan;87(1):e13511. doi: 10.1111/aji.13511. Epub 2021 Dec 4. PMID 34738274
- [Background] Brosens I, Pijnenborg R, Vercruysse L, Romero R. The "Great Obstetrical Syndromes" are associated with disorders of deep placentation. Am J Obstet Gynecol. 2011 Mar;204(3):193-201. doi: 10.1016/j.ajog.2010.08.009. Epub 2010 Nov 20. PMID 21094932
- [Background] Bartsch E, Medcalf KE, Park AL, Ray JG; High Risk of Pre-eclampsia Identification Group. Clinical risk factors for pre-eclampsia determined in early pregnancy: systematic review and meta-analysis of large cohort studies. BMJ. 2016 Apr 19;353:i1753. doi: 10.1136/bmj.i1753. PMID 27094586
- [Background] Brennan LJ, Morton JS, Davidge ST. Vascular dysfunction in preeclampsia. Microcirculation. 2014 Jan;21(1):4-14. doi: 10.1111/micc.12079. PMID 23890192
- [Background] Mayrink J, Souza RT, Feitosa FE, Rocha Filho EA, Leite DF, Vettorazzi J, Calderon IM, Sousa MH, Costa ML, Baker PN, Cecatti JG; Preterm SAMBA study group. Incidence and risk factors for Preeclampsia in a cohort of healthy nulliparous pregnant women: a nested case-control study. Sci Rep. 2019 Jul 2;9(1):9517. doi: 10.1038/s41598-019-46011-3. PMID 31266984
- [Background] Berntsen S, Larsen EC, la Cour Freiesleben N, Pinborg A. Pregnancy outcomes following oocyte donation. Best Pract Res Clin Obstet Gynaecol. 2021 Jan;70:81-91. doi: 10.1016/j.bpobgyn.2020.07.008. Epub 2020 Jul 15. PMID 32741624
- [Background] Preaubert L, Vincent-Rohfritsch A, Santulli P, Gayet V, Goffinet F, Le Ray C. Outcomes of pregnancies achieved by double gamete donation: A comparison with pregnancies obtained by oocyte donation alone. Eur J Obstet Gynecol Reprod Biol. 2018 Mar;222:1-6. doi: 10.1016/j.ejogrb.2017.12.026. Epub 2017 Dec 15. PMID 29309921
- [Background] Nejdet S, Bergh C, Kallen K, Wennerholm UB, Thurin-Kjellberg A. High risks of maternal and perinatal complications in singletons born after oocyte donation. Acta Obstet Gynecol Scand. 2016 Aug;95(8):879-86. doi: 10.1111/aogs.12904. Epub 2016 Apr 28. PMID 27060438
- [Background] Rodriguez-Wallberg KA, Berger AS, Fagerberg A, Olofsson JI, Scherman-Pukk C, Lindqvist PG, Nasiell J. Increased incidence of obstetric and perinatal complications in pregnancies achieved using donor oocytes and single embryo transfer in young and healthy women. A prospective hospital-based matched cohort study. Gynecol Endocrinol. 2019 Apr;35(4):314-319. doi: 10.1080/09513590.2018.1528577. Epub 2019 Jan 9. PMID 30626251
- [Background] Storgaard M, Loft A, Bergh C, Wennerholm UB, Soderstrom-Anttila V, Romundstad LB, Aittomaki K, Oldereid N, Forman J, Pinborg A. Obstetric and neonatal complications in pregnancies conceived after oocyte donation: a systematic review and meta-analysis. BJOG. 2017 Mar;124(4):561-572. doi: 10.1111/1471-0528.14257. Epub 2016 Sep 5. PMID 27592694
- [Background] Serhal PF, Craft IL. Oocyte donation in 61 patients. Lancet. 1989 May 27;1(8648):1185-7. doi: 10.1016/s0140-6736(89)92762-1. PMID 2566746
- [Background] Hogan RG, Wang AY, Li Z, Hammarberg K, Johnson L, Mol BW, Sullivan EA. Oocyte donor age has a significant impact on oocyte recipients' cumulative live-birth rate: a population-based cohort study. Fertil Steril. 2019 Oct;112(4):724-730. doi: 10.1016/j.fertnstert.2019.05.012. Epub 2019 Jun 24. PMID 31248619
- [Background] Wang YA, Farquhar C, Sullivan EA. Donor age is a major determinant of success of oocyte donation/recipient programme. Hum Reprod. 2012 Jan;27(1):118-25. doi: 10.1093/humrep/der359. Epub 2011 Nov 2. PMID 22048992
- [Background] Ginsburg ES, George JS. Older but not wiser: the impact of increasing paternal age on donor oocyte recipient success. Fertil Steril. 2021 Aug;116(2):337-338. doi: 10.1016/j.fertnstert.2021.06.031. Epub 2021 Jul 10. No abstract available. PMID 34253325
- [Background] Lutjen P, Trounson A, Leeton J, Findlay J, Wood C, Renou P. The establishment and maintenance of pregnancy using in vitro fertilization and embryo donation in a patient with primary ovarian failure. Nature. 1984 Jan 12-18;307(5947):174-5. doi: 10.1038/307174a0. PMID 6690997
- [Background] Matthews TJ, Hamilton BE. Delayed childbearing: more women are having their first child later in life. NCHS Data Brief. 2009 Aug;(21):1-8. PMID 19674536
- See also: Webpage for the Danish Society for Fertility Treatment — https://fertilitetsselskab.dk/
- See also: Danish Society For Obstetricians and Gynecologists, guideline on pregnancy after oocyte donation — https://www.dsog.dk/obstetrik

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT07263490/Prot_SAP_000.pdf